CLINICAL TRIAL: NCT00666731
Title: Development and Implementation of The Breast Cancer Collaborative Registry (BCCR)
Brief Title: Breast Cancer Registry for Participants With Breast Cancer or Characteristics of Hereditary Breast Cancer
Acronym: BCCR
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0311-06-EP; P30CA036727 (NIH)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Precancerous Condition
Keywords: male breast cancer; breast cancer; ductal breast carcinoma in situ; lobular breast carcinoma in situ; atypical ductal breast hyperplasia
MeSH Terms: conditions — Breast Neoplasms; Precancerous Conditions; Breast Neoplasms, Male; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical chart review — Demographic information (like address and birth date), the results of physical exams, blood tests, x-rays and other diagnostic and medical procedures and treatments, as well as medical and surgical history.
Other: questionnaire administration — Collection of personal information, medical history, diet and lifestyle habits, any past or current environmental exposures and to re-create a family tree for any cancers that have occurred in any family members. In accordance with OPRR guidelines, no identifying information such as name, address, or date of birth will be used for relatives, but the affected status (cancer, age of onset, year of birth, age of death) will be recorded.
Other: study of socioeconomic and demographic variables — Repository
Procedure: Excess human biological tissue — Tissue procurement.
Procedure: quality-of-life assessment — Cancer care.

SUMMARY:
RATIONALE: Gathering information about patients with breast cancer and their families may help the study of breast cancer in the future.

PURPOSE: This clinical trial is gathering information about patients with breast cancer and their families.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a web-based Breast Cancer Collaborative Registry (BCCR) as a repository for socio-demographic, environmental, clinical history, family history, and biospecimen data collected at the National Comprehensive Cancer Network (NCCN) centers for participants with a personal history of breast cancer and/or characteristics of hereditary breast cancer.
* To merge the data already being collected on breast cancer patients under the Adult Oncology Data Collection Study and newly diagnosed breast cancer patients participating in the NCCN Data Coordinating study at UNMC/NMC.
* To standardize clinical, environmental, socio-demographic, and family history data for breast cancer-related information to be collected and shared for research purposes by Eppley Breast Cancer Research Group breast cancer research collaborators.
* To collect, validate, and disseminate the breast cancer-related data to establish a high-risk cohort for future research into the molecular and biological bases of breast cancer susceptibility and interventional trials.

OUTLINE: This is a multicenter study.

Study participants undergo data collection related to breast cancer studies at one of the National Comprehensive Cancer Network (NCCN) centers for inclusion in the Breast Cancer Collaborative Registry (BCCR). The BCCR is a comprehensive computerized database that serves as a repository for socio-demographic, environmental, clinical history, family history, and biospecimen data collected for breast cancer patients treated on UNMC protocols. Central features of the registry include standardized data-entry forms and a relational database that can be used as a resource for the study of the pathology, immunology, cytogenetics, molecular biology, epidemiology, clinical features, and outcome of patients with benign, pre-malignant, or malignant breast disease.

Study participants complete a self-administered electronic or paper-based survey and a medical history questionnaire at baseline to provide information on demographics (e.g., age and sex); personal and family medical history; treatment history; lifestyle, physical activity, and dietary habits; quality of life; environmental exposure history; and the family tree for inclusion in the registry. Participants also undergo telephone or in-person structured interviews conducted by study coordinators, genetic counselors, or the System Coordinator of the BCCR to provide additional information or clarification of the information provided in the questionnaires.

Study participants also undergo review of their medical records and pathology reports to obtain detailed medical and treatment-related information for inclusion in the registry. The information collected includes retrospective and prospective disease-specific data (e.g., diagnosis, grade/stage, and laboratory values) and longitudinal outcome data (e.g., response to treatment, toxicity, survival, relapse) derived during prospective clinical follow-up.

Study participants are followed periodically to update relevant health and family histories.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis or history of breast cancer
* Atypical hyperplasia
* Ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) as defined in the National Comprehensive Cancer Network Breast and/or Ovarian Genetic Assessment Guidelines, v.1.2006
* Characteristics of hereditary breast cancer, as defined in the National Comprehensive Cancer Network Breast and/or Ovarian Genetic Assessment Guidelines, v.1.2006 (relatives have been diagnosed with breast and/or ovarian cancer) OR have a breast cancer risk of > 1.67% over 5 years as estimated by the GAIL Model

Exclusion Criteria:

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adult individuals (male and female) who have a personal diagnosis/history of breast cancer, atypical hyperplasia, ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) (as stated in the NCCN Breast and/or Ovarian Genetic Assessment Guidelines v.1.2006 (Appendix A)
  2. Adult individuals who have characteristics of hereditary breast cancer, as defined in the NCCN Breast and/or Ovarian Genetic Assessment Guidelines v.1.2006 (Appendix A) or who have a breast cancer risk of > 1.67% over 5 years as estimated by GAIL Model (Appendix C )
  3. Age 19 or greater
  4. Able to provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 4945 (Actual)
Dates: Start 2006-10-12 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

PRIMARY OUTCOMES:
Implementation of a web-based Breast Cancer Collaborative Registry at the National Comprehensive Cancer Network (NCCN) centers | Ongoing
  Web-based registry
Merger of data collected under the Adult Oncology Data Collection Study and the National Comprehensive Cancer Network Data Coordinating study at UNMC/NMC | Ongoing
  Web-based registries.
Standardization of clinical, environmental, socio-demographic, and family history data collected for breast cancer-related research and shared by the Eppley Breast Cancer Research Group collaborators | Ongoing
  Web-based registry.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Cowan, MD, PhD, Principal Investigator — University of Nebraska
Locations (65):
- United States (65):
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Centura - Porter Adventist Hospital, Denver, Colorado
  - Centura - St. Anthony Hospital, Lakewood, Colorado
  - Centura - Parker Adventist Hospital, Parker, Colorado
  - Centura - St. Mary Corwin Medical Center, Pueblo, Colorado
  - Halifax Health Medical Center, Daytona Beach, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Hlaifax Health Medical Center, Daytona Beach, Florida
  - Florida Hospital Deland, DeLand, Florida
  - Florida Hospital FISH, Orange City, Florida
  - Halifax Health Medical Center, Ormond Beach, Florida
  - Florida Hospital Flagler, Palm Coast, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Community Cancer Care, Anderson, Indiana
  - Community Clinical Research Center, Anderson, Indiana
  - Community Hospital of Anderson and Madison County, Inc, Anderson, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Genesis Medical Center, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Mercy Medical Center, North Iowa, Mason City, Iowa
  - Abben Cancer Center, Spencer, Iowa
  - Covenant Medical Center, Inc, Waterloo, Iowa
  - Saint Luke's Cancer Instititue, South, Overland Park, Kansas
  - Tulane University, New Orleans, Louisiana
  - Central Maine Medical Center, Bennett Breast Care Center, Lewiston, Maine
  - Central Maine Medical Center, Cynthia A. Rydhom Cancer Treatment Center, Lewiston, Maine
  - Central Maine Medical Center, Hematology Oncology Associates, Lewiston, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Research Associates, Lewiston, Maine
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - William E Kahlert Regional Cancer Center, Westminster, Maryland
  - Holyoke Medical Center, Holyoke, Massachusetts
  - Beth Israel Deaconess Hospital, Plymouth, Massachusetts
  - Mercy Hospital - Joplin, Joplin, Missouri
  - Saint Luke's Cancer Institute - East, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Cancer Institute - Kansas City North, Kansas City, Missouri
  - Saint Luke's Cancer Institute - Liberty, Liberty, Missouri
  - Heartland Regional Medical Center dba Mosaic Life Care, Saint Joseph, Missouri
  - Heartland Regional Medical Center dba Cancer Care, St. Joseph, Mosaic Life Care, Saint Joseph, Missouri
  - Mary Lanning Healthcare/Morrison Cancer Center, Hastings, Nebraska
  - Good Samaritan Hospital/Cancer Center, Kearney, Nebraska
  - Faith Regional Health Services, Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska
  - Regional West Health Services, Scottsbluff, Nebraska
  - C.R. Wood Cancer Center, Glens Falls Hospital, Glens Falls, New York
  - Faxton St. Lukes (St. Elizabeth campus), Utica, New York
  - Faxton St. Luke's Healthcare (Mohawk Valley Health Systems), Utica, New York
  - Faxton St. Luke's Healthcare (St. Luke's Campus), Utica, New York
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Trinity Hospital Cancer Care Center, Minot, North Dakota
  - Avera Medical Group Oncology and Hematology Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute, Mitchell, South Dakota
  - Avera Cancer Center, Sioux Falls, South Dakota
  - Rutland Regional Medical Center, Rutland, Vermont
  - Wheaton Franciscan Healthcare - Elmbrook Memorial Hospital, Brookfield, Wisconsin
  - Wheaton Franciscan Healthcare - Reiman Cancer Care, Franklin, Wisconsin
  - Wheaton Franciscan Healthcare - All Saints, Racine, Wisconsin
  - Wheaton Franciscan Healthcare - Wauwatosa Cancer Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No